CLINICAL TRIAL: NCT05789069
Title: A Phase 1a/1b, Open-Label, Multi-Center, Dose Escalation and Expansion Study of HFB200603 (Anti-BTLA Antibody) as a Single Agent and in Combination With Tislelizumab (Anti-PD-1 Antibody) in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of HFB200603 as a Single Agent and in Combination With Tislelizumab in Adult Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HiFiBiO Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HFB-200603-01; 2022-502891-22-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-24; First posted 2023-03-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma; Melanoma; Non Small Cell Lung Cancer; Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Colorectal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation - HFB200603 monotherapy (Experimental): Participants will be administered HFB200603 at dose levels 1-4 as an intravenous infusion to determine the Recommended Dose for Expansion (RDE).
  Interventions: Drug: HFB200603
- Dose Escalation - HFB200603 in combination with tislelizumab (Experimental): Participants will be administered HFB200603 at dose levels 1-3 in combination with one dose level of tislelizumab as an intravenous infusion to determine the combination Recommended Doses for Expansion (RDEs).
  Interventions: Drug: HFB200603; Drug: Tislelizumab
- Dose Expansion - HFB200603 monotherapy (optional) (Experimental): Participants will be administered HFB200603 at monotherapy RDE as an intravenous infusion.
  Interventions: Drug: HFB200603
- Dose Expansion - HFB200603 in combination with tislelizumab (Experimental): Participants will be administered HFB200603 in combination with tislelizumab at combination RDEs as an intravenous infusion. Based on the cancer type, participants will be randomized to combination HFB200603 RDE 1 or RDE 2.
  Interventions: Drug: HFB200603; Drug: Tislelizumab

INTERVENTIONS:
Drug: HFB200603 — Participants will be administered HFB200603 as described in the experimental arm.
Drug: Tislelizumab — Participants will be administered tislelizumab as described in the experimental arm.
  Other Names: BGB-A317
  Arms: Dose Escalation - HFB200603 in combination with tislelizumab; Dose Expansion - HFB200603 in combination with tislelizumab

SUMMARY:
The purpose of this study is to test the safety and tolerability of HFB200603 as a single agent and in combination with tislelizumab in patients with advanced cancers. There are two parts in this study. During the escalation part, groups of participants will receive increasing doses of HFB200603 as a monotherapy or in combination with tislelizumab until a safe and tolerable dose of HFB200603 as a single agent or combination therapy is determined. During the expansion part, participants will take the doses of HFB200603 as a monotherapy (optional arm) or in combination with tislelizumab that were determined from the escalation part of the study and will be assigned to a group based on the type of cancer the participants have.

DETAILED DESCRIPTION:
This is a Phase 1a/b, first in human, open-label, dose escalation and expansion study in adults with advanced cancers. The study will comprise of

1. A Screening Period of up to 28 days
2. A Treatment Period during which participants will receive the study drug on the first day of each cycle where each cycle is 21 days. Number of cycles depends on how the disease responds to the study drug
3. A Follow-up Period which involves 2 visits

ELIGIBILITY:
Inclusion Criteria:

* Patient must have one of the following cancers and previously received the following lines of systemic therapy for the advanced/metastatic disease:

  * Renal cell carcinoma: at least 2 lines of therapy
  * Non-small cell lung cancer: at least 2 lines of therapy
  * Melanoma:

    * BRAF V600E positive: must have received at least 2 lines of therapy
    * BRAF V600E negative: must have received at least 1 line of therapy
  * Gastric cancer: at least 1 line of therapy
  * Colorectal cancer: at least 3 lines of therapy
* Suitable site to biopsy at pre-treatment and on-treatment
* Measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group performance status of 0 or 1

Exclusion Criteria:

* Systemic anti-cancer therapy within 2 weeks prior to start of study drug or within 4 weeks for immune-oncologic therapy. For cytotoxic agents with major delayed toxicity (e.g., mitomycin C), 6 weeks of washout are mandated.
* Therapeutic radiation therapy within the past 2 weeks
* Active autoimmune diseases or history of autoimmune disease that may relapse
* Any malignancy ≤ 5 years before first dose of study drug except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively
* Systemic steroid therapy (>10 mg/day of prednisone or equivalent) or any immune suppressive medication ≤ 14 days before first dose
* Patients with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or stabilized, except for adverse events not considered a likely safety risk (e.g., alopecia, neuropathy, and specific laboratory abnormalities)
* Severe or unstable medical condition, including uncontrolled diabetes, coagulopathy, or unstable psychiatric condition
* Major surgery within 28 days of the first dose of study drug
* History of interstitial lung disease, non-infectious pneumonitis, or uncontrolled lung diseases including pulmonary fibrosis or acute lung diseases. For combination only: non-small cell lung cancer patients, or patients with significantly impaired pulmonary function or who require supplemental oxygen at baseline must undergo an assessment of pulmonary function at screening
* History of allergic reactions, immune related reactions, or cytokine release syndrome (CRS) attributed to compounds of similar chemical or biologic composition to monoclonal antibodies or any excipient of HFB200603 or tislelizumab
* For combination only: Prior randomization in a tislelizumab study regardless of the treatment arm, until the primary and key secondary endpoints of the study have read out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) meeting protocol-defined Dose-Limiting Toxicity (DLT) criteria during Dose Escalation | The first cycle of treatment (Day 1 up to Day 21)
  Severity of adverse events will be based on common terminology criteria for adverse events (CTCAE) version 5.0
Number of participants with AEs | Cycle 1 Day 1 to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years
  Severity of AEs will be assessed based on CTCAE version 5.0 (except for cytokine release syndrome which will be assessed by American Society for Transplantation and Cellular Therapy grading)
Number of participants with changes in laboratory values | Cycle 1 Day 1 to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years
Number of participants with changes in vital signs | Cycle 1 Day 1 to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years
Number of participants with changes in electrocardiogram (ECG) | Cycle 1 Day 1 to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years
Number of participants with changes in tolerability (dose interruptions and dose intensity) | Cycle 1 Day 1 to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years
To determine a Recommended Phase 2 Dose (RP2D) during Dose Expansion | Cycle 1 Day 1 to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-RECIST (iRECIST) | Baseline to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years
Disease Control Rate (DCR) as determined by RECIST 1.1 and iRECIST | Baseline to 90 days after the last dose of study drug(s) (each cycle is 21 days), assessed up to 3 years
Duration of Response (DOR) as determined by RECIST 1.1 and iRECIST | Start of first response to first date of disease progression, clinical progression or death, whichever occurs first, assessed up to 3 years
Progression Free Survival (PFS) as determined by RECIST 1.1 and iRECIST | Baseline to disease progression or death, whichever occurs first, assessed up to 3 years
Minimum serum concentration (Cmin) | Cycle 1 Day 1 to day of the last dose of study drug(s) (each cycle is 21 days), through study completion, an average of 3 year
Maximum serum concentration (Cmax) | Cycle 1 Day 1 to day of the last dose of study drug(s) (each cycle is 21 days), through study completion, an average of 3 year
Area under the concentration versus time curve (AUC) | Cycle 1 Day 1 to day of the last dose of study drug(s) (each cycle is 21 days), through study completion, an average of 3 year
Terminal half-life (T1/2) | Cycle 1 Day 1 to day of the last dose of study drug(s) (each cycle is 21 days), through study completion, an average of 3 year
Serum concentration for measurement of anti-HFB200603 antibodies | Cycle 1 Day 1 to day of the last dose of study drug(s) (each cycle is 21 days), through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - New Experimental Therapeutics of Virginia - NEXT Oncology, Fairfax, Virginia
- Italy (3):
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - UOC Fase I - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Spain (5):
  - Clinica Universidad de Navarra - Madrid, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - CIOCC, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia